CLINICAL TRIAL: NCT00803049
Title: Long-term Extension of the Multinational, Double-blind, Placebo Controlled Study EFC6049 (HMR1726D/3001) to Document the Safety of Two Doses of Teriflunomide (7 and 14 mg) in Patients With Multiple Sclerosis With Relapses
Brief Title: Long Term Safety and Efficacy Study of Teriflunomide 7 mg or 14 mg in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTS6050; 2006-003361-14 (EudraCT Number)
Record Dates: First submitted 2008-12-01; First posted 2008-12-05 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Oral treatment
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo/Teriflunomide 7 mg (Experimental): Participants who completed treatment of placebo (for teriflunomide) tablet once daily (QD) for 108 weeks in EFC6049 study, received teriflunomide tablet 7 mg QD for 288 weeks in this extension study.
  Interventions: Drug: Teriflunomide (HMR1726)
- Teriflunomide 7 mg/7 mg (Experimental): Participants who completed treatment of teriflunomide 7 mg tablet QD for 108 weeks in EFC6049 study, continued their treatment with teriflunomide 7 mg tablet QD for 288 weeks in this extension study.
  Interventions: Drug: Teriflunomide (HMR1726)
- Placebo/Teriflunomide 14 mg (Experimental): Participants who completed treatment of placebo (for teriflunomide) tablet QD for 108 weeks in EFC6049, study received teriflunomide 14 mg tablet QD for 288 weeks in this extension study.
  Interventions: Drug: Teriflunomide (HMR1726)
- Teriflunomide 14 mg/14 mg (Experimental): Participants who completed treatment of teriflunomide 14 mg tablet QD for 108 weeks in EFC6049 study, continued their treatment with teriflunomide 14 mg tablet QD for 288 weeks in this extension study.
  Interventions: Drug: Teriflunomide (HMR1726)

INTERVENTIONS:
Drug: Teriflunomide (HMR1726) — Tablet, oral administration QD.
  Other Names: Aubagio

SUMMARY:
The primary objective of this study was to document the long-term safety and tolerability of teriflunomide in Multiple Sclerosis (MS) participants with relapse.

The secondary objective was to document the long-term efficacy on disability progression, relapse rate and Magnetic Resonance Imaging (MRI) parameters.

DETAILED DESCRIPTION:
Participants completing the EFC6049 (HMR1726D/3001) study were given the opportunity to continue in the extension study;

* participants receiving teriflunomide 7 mg or 14 mg were blindly maintained on the same dose of teriflunomide.
* participants receiving placebo were randomized at a 1:1 ratio to teriflunomide 7 mg or 14 mg.

The study period per participant was broken down as follows:

* Double-blind treatment: up to a maximum of 288 weeks or until teriflunomide was commercially available in the country where participant lived,
* Post-washout follow-up: 4 weeks after last treatment intake. No post-washout follow up if participant continued on teriflunomide treatment by obtaining its commercial form after end of the study.

The total duration of the extension was 292 weeks (about 6 years) from the first participant enrolled or until teriflunomide is commercially available in the country where participant lived.

ELIGIBILITY:
Inclusion Criteria:

* Participant who completed the previous double-blind placebo-controlled study EFC6049 and who did not meet criteria for treatment withdrawal.
* Willingness to participate in a long-term safety/efficacy trial.

Exclusion Criteria:

* Any known condition or circumstance that would prevent in the investigator's opinion, compliance or completion of the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 742 (Actual)
Dates: Start 2006-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (116):
- United States (4):
  - Investigational Site Number 1032, Maitland, Florida
  - Investigational Site Number 1038, Fort Wayne, Indiana
  - Investigational Site Number 1033, Detroit, Michigan
  - Investigational Site Number 1037, Allentown, Pennsylvania
- Austria (4):
  - Investigational Site Number 1603, Graz
  - Investigational Site Number 1604, Innsbruck
  - Investigational Site Number 1601, Vienna
  - Investigational Site Number 1602, Vienna
- Canada (12):
  - Investigational Site Number 1208, Calgary
  - Investigational Site Number 1212, Gatineau
  - Investigational Site Number 1205, Greenfield Park
  - Investigational Site Number 1201, Halifax
  - Investigational Site Number 1206, London
  - Investigational Site Number 1203, Montreal
  - Investigational Site Number 1204, Ottawa
  - Investigational Site Number 1202, Québec
  - Investigational Site Number 1211, St. John's
  - Investigational Site Number 1209, Toronto
  - Investigational Site Number 1210, Vancouver
  - Investigational Site Number 1207, Winnipeg
- Chile (5):
  - Investigational Site Number 3804, Santiago
  - Investigational Site Number 3802, Santiago
  - Investigational Site Number 3803, Santiago
  - Investigational Site Number 3801, Santiago
  - Investigational Site Number 3805, Viña del Mar
- Investigational Site Number 4101, Olomouc, Czechia
- Denmark (3):
  - Investigational Site Number 4801, Glostrup Municipality
  - Investigational Site Number 4804, Sønderborg
  - Investigational Site Number 4802, Vejle
- Estonia (2):
  - Investigational Site Number 1502, Tallinn
  - Investigational Site Number 1501, Tartu
- Finland (4):
  - Investigational Site Number 2203, Helsinki
  - Investigational Site Number 2206, Pori
  - Investigational Site Number 2201, Tampere
  - Investigational Site Number 2202, Turku
- France (14):
  - Investigational Site Number 2415, Besançon
  - Investigational Site Number 2403, Clermont-Ferrand
  - Investigational Site Number 2408, Dijon
  - Investigational Site Number 2413, Lille
  - Investigational Site Number 2404, Limoges
  - Investigational Site Number 2401, Lyon
  - Investigational Site Number 2409, Marseille
  - Investigational Site Number 2402, Montpellier
  - Investigational Site Number 2405, Nancy
  - Investigational Site Number 2414, Nantes
  - Investigational Site Number 2407, Nice
  - Investigational Site Number 2410, Paris
  - Investigational Site Number 2406, Rennes
  - Investigational Site Number 2411, Toulouse
- Germany (11):
  - Investigational Site Number 2011, Berlin
  - Investigational Site Number 2001, Berlin
  - Investigational Site Number 2000, Bochum
  - Investigational Site Number 2012, Erbach im Odenwald
  - Investigational Site Number 2004, Essen
  - Investigational Site Number 2005, Giessen
  - Investigational Site Number 2007, Hanover
  - Investigational Site Number 2008, Münster
  - Investigational Site Number 2010, Offenbach
  - Investigational Site Number 2009, Rostock
  - Investigational Site Number 2003, Wiesbaden
- Italy (9):
  - Investigational Site Number 2819, Bari
  - Investigational Site Number 2827, Fidenza
  - Investigational Site Number 2803, Florence
  - Investigational Site Number 2814, Gallarate
  - Investigational Site Number 2808, Milan
  - Investigational Site Number 2812, Padua
  - Investigational Site Number 2809, Pavia
  - Investigational Site Number 2813, Roma
  - Investigational Site Number 2824, Roma
- Netherlands (4):
  - Investigational Site Number 4602, 's-Hertogenbosch
  - Investigational Site Number 4605, Breda
  - Investigational Site Number 4601, Nijmegen
  - Investigational Site Number 4604, Sittard-Geleen
- Norway (2):
  - Investigational Site Number 3601, Oslo
  - Investigational Site Number 3604, Tønsberg
- Poland (9):
  - Investigational Site Number 3008, Bialystok
  - Investigational Site Number 3009, Bialystok
  - Investigational Site Number 3007, Gdansk
  - Investigational Site Number 3005, Lodz
  - Investigational Site Number 3006, Lublin
  - Investigational Site Number 3004, Lublin
  - Investigational Site Number 3001, Poznan
  - Investigational Site Number 3002, Warsaw
  - Investigational Site Number 3003, Warsaw
- Portugal (2):
  - Investigational Site Number 4201, Coimbra
  - Investigational Site Number 4203, Lisbon
- Russia (7):
  - Investigational Site Number 3203, Moscow
  - Investigational Site Number 3205, Moscow
  - Investigational Site Number 3207, Nizhny Novgorod
  - Investigational Site Number 3208, Novosibirsk
  - Investigational Site Number 3201, Saint Petersburg
  - Investigational Site Number 3202, Saint Petersburg
  - Investigational Site Number 3206, Saint Petersburg
- Investigational Site Number 3401, Stockholm, Sweden
- Investigational Site Number 1802, Basel, Switzerland
- Turkey (Türkiye) (4):
  - Investigational Site Number 5003, Izmir
  - Investigational Site Number 5006, Izmir
  - Investigational Site Number 5005, Kocaeli
  - Investigational Site Number 5001, Sihhiye / Ankara
- Ukraine (9):
  - Investigational Site Number 3504, Dnipropetrovsk
  - Investigational Site Number 3505, Ivano-Frankivsk
  - Investigational Site Number 3506, Kharkiv
  - Investigational Site Number 3510, Kharkiv
  - Investigational Site Number 3508, Lviv
  - Investigational Site Number 3502, Odesa
  - Investigational Site Number 3509, Uzhhorod
  - Investigational Site Number 3507, Vinnitsa
  - Investigational Site Number 3501, Zaporizhzhya
- United Kingdom (8):
  - Investigational Site Number 2604, Dundee
  - Investigational Site Number 2607, London
  - Investigational Site Number 2608, London
  - Investigational Site Number 2600, Newcastle upon Tyne
  - Investigational Site Number 2601, Nottingham
  - Investigational Site Number 2609, Plymouth
  - Investigational Site Number 2606, Sheffield
  - Investigational Site Number 2602, Stoke-on-Trent

REFERENCES:
- [Derived] Sprenger T, Kappos L, Sormani MP, Miller AE, Poole EM, Cavalier S, Wuerfel J. Effects of teriflunomide treatment on cognitive performance and brain volume in patients with relapsing multiple sclerosis: Post hoc analysis of the TEMSO core and extension studies. Mult Scler. 2022 Oct;28(11):1719-1728. doi: 10.1177/13524585221089534. Epub 2022 Apr 29. PMID 35485424
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488
- [Derived] Sprenger T, Kappos L, Radue EW, Gaetano L, Mueller-Lenke N, Wuerfel J, Poole EM, Cavalier S. Association of brain volume loss and long-term disability outcomes in patients with multiple sclerosis treated with teriflunomide. Mult Scler. 2020 Sep;26(10):1207-1216. doi: 10.1177/1352458519855722. Epub 2019 Jun 14. PMID 31198103
- [Derived] Sormani MP, Truffinet P, Thangavelu K, Rufi P, Simonson C, De Stefano N. Predicting long-term disability outcomes in patients with MS treated with teriflunomide in TEMSO. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 28;4(5):e379. doi: 10.1212/NXI.0000000000000379. eCollection 2017 Sep. PMID 28680917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 117 centres in 21 countries between 16 October 2006 and 23 December 2015. A total of 742 participants who completed study EFC6049 (NCT00134563), entered in this extension study (LTS6050 [NCT00803049]).
Pre-assignment Details: Participants who received placebo in EFC6049 study were randomized in 1:1 ratio to receive either teriflunomide 7 mg/day or 14 mg/day and, those who received teriflunomide 7 mg/day or 14 mg/day in EFC6049 (NCT00134563) received same double-blind treatment in this extension study.
Period: Overall Study
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Started | 129 (Randomized in extension study) | 252 (Randomized in extension study) | 108 (Randomized in extension study) | 253 (Randomized in extension study)
Treated | 129 | 252 | 108 | 251
Safety Population | 129 | 254 (Included 1 participant from Placebo/Teriflunomide 14 mg and 1 from Teriflunomide14 mg/14 mg arm) | 107 (1 participant received Teriflunomide 7 mg and analysed in Teriflunomide 7 mg/7 mg arm) | 250 (1 participant received Teriflunomide 7 mg and analysed in Teriflunomide 7 mg/7 mg arm)
Completed | 68 | 134 | 64 | 151
Not Completed | 61 | 118 | 44 | 102
Not completed — Adverse Event | 21 | 33 | 13 | 27
Not completed — Lack of Efficacy | 10 | 19 | 6 | 13
Not completed — Lost to Follow-up | 0 | 2 | 0 | 3
Not completed — Death | 2 | 1 | 0 | 2
Not completed — Progressive Disease | 6 | 10 | 6 | 6
Not completed — Withdrawal by Subject | 19 | 43 | 16 | 44
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Randomized and Not Treated | 0 | 0 | 0 | 2
Not completed — Other than Specified Above | 3 | 9 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg | Total
Number analyzed (Participants) | 129 | 252 | 108 | 253 | 742
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (8.5) | 38.0 (8.8) | 37.6 (8.5) | 38.6 (8.4) | 38.4 (8.6)
Gender [Count of Participants; unit: Participants]
  Female | 94 | 175 | 85 | 182 | 536
  Male | 35 | 77 | 23 | 71 | 206

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received investigational medicinal product (IMP) without regard to possibility of causal relationship with this treatment. TEAEs: AEs that developed or worsened or became serious during on-treatment period which was defined as the period from the time of first dose of study drug (in LTS6050) up to 4 weeks (28 days) after last dose of study drug. Serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included both serious and non-serious AEs.
Time Frame: Baseline (LTS6050) up to 28 days after last dose of study drug up to 450 weeks
Population: Safety population: all participants randomized in the LTS6050 study and exposed to IMP during the LTS6050 study treatment period, regardless of the amount of treatment administered. The safety analysis was conducted as the treatment received.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Teriflunomide 7 mg: Participants who completed treatment of placebo (for teriflunomide) tablet QD for 108 weeks in EFC6049 study, received teriflunomide tablet 7 mg QD for 288 weeks in this extension study.
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 129 | 254 | 107 | 250
percentage of participants
  Any TEAE | 93.8 | 91.3 | 94.4 | 91.2
  Any Treatment Emergent SAE | 24.8 | 28.0 | 21.5 | 24.8
  Any TEAE Leading to Death | 2.3 | 0.8 | 0 | 0.8
  Any TEAE Leading to Permanent Discontinuation | 17.1 | 12.2 | 12.1 | 10.8

2. Secondary Outcome: Time to 12 Week Sustained Disability Progression (DP): Kaplan-Meier Estimates of the Rate of DP
Description: Sustained DP defined as sustained increase of at least 1 point from baseline (EFC6049) expanded disability status scale (EDSS) score (0.5 point for participants with baseline EDSS>5.5) persisting for at least 12 weeks. EDSS: an ordinal scale qualifies disability in participants with MS. EDSS total score range: 0 (normal neurological examination) to 10 (death due to Multiple Sclerosis [MS]). Probability of DP at 12 weeks was estimated using Kaplan-Meier method on time to DP defined as date of first DP minus (-) date of randomization in EFC6049 study +1 day. Participants free of DP (no DP observed on treatment) were censored at the date of last on-treatment EDSS evaluation in LTS6050. Kaplan-Meier method consists in computing probabilities of non-occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t.
Time Frame: Up to 10.8 years (EFC6049: 108 weeks + LTS6050: 450 weeks)
Population: Intent-to-treat (ITT) (EFC6049+ LTS6050) population: all participants randomized in both EFC6049 and LTS6050 studies that had at least 1-day IMP exposure during both EFC6049 and LTS6050 studies. Analysis for this outcome measure was performed on the combined data of EFC6049 andLTS6050 study, as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 129 | 252 | 108 | 251
Probability | 0.544 [0.441 to 0.646] | 0.494 [0.423 to 0.565] | 0.627 [0.444 to 0.811] | 0.473 [0.403 to 0.543]
Statistical Analysis 1: Comparison: Placebo/Teriflunomide 7 mg vs Teriflunomide 7 mg/7 mg; Analysis was performed using Log-rank test with treatment, EDSS strata at baseline and region as covariates. Estimation was performed using Cox proportional hazard model with treatment, EDSS strata at baseline and region as covariates; Test type: Superiority or Other; p = 0.2079, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.824, 95% CI 2-sided [0.602 to 1.128] — Placebo/Teriflunomide 7 mg vs. Teriflunomide 7 mg/7 mg
Statistical Analysis 2: Comparison: Placebo/Teriflunomide 14 mg vs Teriflunomide 14 mg/14 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3039, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.825, 95% CI 2-sided [0.591 to 1.152] — Placebo/Teriflunomide 14 mg vs.Teriflunomide 14 mg/14 mg
Statistical Analysis 3: Comparison: Teriflunomide 7 mg/7 mg vs Teriflunomide 14 mg/14 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8271, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.963, 95% CI 2-sided [0.736 to 1.260] — Teriflunomide 7 mg/7 mg vs. Teriflunomide 14 mg/14 mg

3. Secondary Outcome: Time to 24 Week Sustained Disability Progression (DP): Kaplan-Meier Estimates of the Rate of DP
Description: Sustained DP was defined as sustained increase of at least 1 point from baseline (EFC6049) EDSS score (0.5 point for participants with baseline EDSS>5.5) persisting for at least 24 weeks. EDSS: an ordinal scale qualifies disability in participants with MS. EDSS total score range: 0 (normal neurological examination) to 10 (death due to MS). Probability of DP at 24 weeks was estimated using Kaplan-Meier method on time to DP defined as date of first DP minus (-) date of randomization in EFC6049 study +1 day. Participants free of DP (no DP observed on treatment) were censored at the date of last on-treatment EDSS evaluation in LTS6050. Kaplan-Meier method consists in computing probabilities of non-occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t.
Time Frame: Up to 10.8 years (EFC6049: 108 weeks + LTS6050: 450 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 129 | 252 | 108 | 251
Probability | 0.444 [0.338 to 0.550] | 0.434 [0.363 to 0.504] | 0.518 [0.411 to 0.624] | 0.438 [0.367 to 0.509]
Statistical Analysis 1: Comparison: Placebo/Teriflunomide 7 mg vs Teriflunomide 7 mg/7 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8017, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.961, 95% CI 2-sided [0.678 to 1.362] — Placebo/Teriflunomide 7 mg vs. Teriflunomide 7 mg/7 mg
Statistical Analysis 2: Comparison: Placebo/Teriflunomide 14 mg vs Teriflunomide 14 mg/14 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1866, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.790, 95% CI 2-sided [0.559 to 1.117] — Placebo/Teriflunomide 14 mg vs. Teriflunomide 14 mg/14 mg
Statistical Analysis 3: Comparison: Teriflunomide 7 mg/7 mg vs Teriflunomide 14 mg/14 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8763, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 1.020, 95% CI 2-sided [0.767 to 1.357] — Teriflunomide 7 mg/7 mg vs. Teriflunomide 14 mg/14 mg

4. Secondary Outcome: Percentage of Participants Free of Sustained Disability Progression (DP)
Description: Sustained DP was defined as sustained increase of at least 1 point from baseline (EFC6049) EDSS score (0.5 point for participants with baseline EDSS>5.5) persisting for at least 12 weeks and 24 weeks. EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder, cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicates worse neurological function. Percentage of participants who were considered as free of disability progression confirmed after 12 week sustained progression and 24 week sustained progression were reported. Analysis for this outcome measure was performed on combined data of EFC6049 and LTS6050 study, as pre-specified in protocol.
Time Frame: Up to 10.8 years since EFC6049 randomization (EFC6049: 108 weeks + LTS6050: 450 weeks)
Population: Intent-to-treat (ITT) (EFC6049 [NCT00134563] + LTS6050) population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 129 | 252 | 108 | 251
percentage of participants
  Free of DP Sustained for 12 Weeks | 45.6 | 50.6 | 37.3 | 52.7
  Free of DP Sustained for 24 Weeks | 55.6 | 56.6 | 48.2 | 56.2

5. Secondary Outcome: Annualized MS Relapse Rate (ARR): Poisson Regression Estimates
Description: ARR was obtained from total number of confirmed relapses that occurred during treatment period divided by sum of treatment durations in LTS6050 study only. Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever was to be confirmed by an increase in EDSS score or Functional System (FS) scores. EDSS: an ordinal scale qualifies disability. EDSS total score range: 0 (normal neurological examination) to 10 (death due to MS). FSS: to assess the neurological function. Total score range: 0 (normal) - 6(worse), higher scores = worse neurological function. To account for the different treatment duration among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log transformed treatment duration as "offset" variable; treatment group, region of enrolment and baseline EDSS stratum as covariates).
Time Frame: Up to 8 years since LTS6050 randomization
Population: ITT(LTS6050) population: all participants who were randomized in the LTS6050 study and had at least 1-day IMP exposure during the LTS6050 study.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 129 | 252 | 108 | 251
relapses per participant-year | 0.216 [0.162 to 0.288] | 0.183 [0.149 to 0.225] | 0.176 [0.132 to 0.236] | 0.160 [0.129 to 0.198]

6. Secondary Outcome: Magnetic Resonance Imaging (MRI) Assessment: Change From Baseline in Total Volume of Abnormal Lesions (Burden of Disease [BOD]) at Week 192 Since LTS6050 Randomization
Description: BOD was assessed by cerebral MRI and defined as the total volume of all abnormal brain tissue (calculated as the sum of the total volume of T2-lesion component and T1-hypointense lesion component).
Time Frame: Baseline, Week 192
Population: ITT (LTS6050 population). Number of participants analyzed=participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: millilitres (ml)
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 49 | 99 | 36 | 103
millilitres (ml) | 5.307 (9.088) | 3.969 (11.135) | 3.720 (6.696) | 3.943 (9.685)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of informed consent form up to 28 days after the last dose of study drug up to Week 450, regardless of seriousness or relationship to investigational product
Description: Reported AEs are TEAEs that is AEs that developed/worsened during the 'on treatment period' (the time from the first dose of study treatment up to 4 weeks [28 days] after the last dose of study treatment). Analysis was performed on safety population and was conducted as per the treatment received.
Groups:
- Teriflunomide 7 mg/7 mg: Participants who completed treatment of teriflunomide 7 mg tablet QD for 108 weeks in EFC6049 study, continued their treatment with teriflunomide 7 mg tablet QD for 288 weeks in this extension study.
  Included 2 participants randomized in placebo and teriflunomide 14 mg arm respectively in EFC6049 study, incorrectly received at least 1 dose of teriflunomide 7 mg. In LTS6050 study, same participants received correct dose of teriflunomide 14 mg but included in Teriflunomide 7mg/7 mg arm for safety analysis.
- Placebo/Teriflunomide 14 mg: Participants who completed treatment of placebo (for teriflunomide) tablet QD for 108 weeks in EFC6049, study received teriflunomide 14 mg tablet QD for 288 weeks in this extension study.
  Excluded 1 participant randomized in placebo arm in EFC6049 study, incorrectly received at least 1 dose of teriflunomide 7 mg. In LTS6050 study, same participant received 14 mg dose but included in teriflunomide 7 mg/7 mg arm for safety analysis.
- Teriflunomide 14 mg/14 mg: Participants who completed treatment of teriflunomide 14 mg tablet QD for 108 weeks in EFC6049 study, continued their treatment with teriflunomide 14 mg tablet QD for 288 weeks in this extension study.
  Excluded 1 participant randomized in 14 mg arm in EFC6049 study, incorrectly received at least 1 dose of teriflunomide 7 mg. In LTS6050 study, same participant received correct dose of 14 mg but included in Teriflunomide 7mg/7 mg arm for safety analysis.
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Serious Adverse Events (participants affected / at risk) | 32/129 | 71/254 | 23/107 | 62/250
Other Adverse Events (participants affected / at risk) | 107/129 | 195/254 | 95/107 | 197/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teriflunomide 7 mg (N=129) | Teriflunomide 7 mg/7 mg (N=254) | Placebo/Teriflunomide 14 mg (N=107) | Teriflunomide 14 mg/14 mg (N=250)
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Uhthoff's phenomenon (Nervous system disorders) | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0 | 0
Facial neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 3 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mesenteric haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Premenstrual cramps (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dolichocolon (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 3 | 6
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Mammoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Osteotomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Miscarriage of partner (Social circumstances) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teriflunomide 7 mg (N=129) | Teriflunomide 7 mg/7 mg (N=254) | Placebo/Teriflunomide 14 mg (N=107) | Teriflunomide 14 mg/14 mg (N=250)
Nasopharyngitis (Infections and infestations) | 34 | 71 | 29 | 81
Influenza (Infections and infestations) | 19 | 39 | 20 | 37
Urinary tract infection (Infections and infestations) | 20 | 31 | 19 | 36
Sinusitis (Infections and infestations) | 7 | 16 | 5 | 28
Upper respiratory tract infection (Infections and infestations) | 15 | 29 | 15 | 28
Bronchitis (Infections and infestations) | 10 | 17 | 9 | 26
Gastroenteritis (Infections and infestations) | 8 | 10 | 8 | 14
Cystitis (Infections and infestations) | 9 | 8 | 4 | 9
Respiratory tract infection (Infections and infestations) | 8 | 10 | 9 | 7
Oral herpes (Infections and infestations) | 3 | 17 | 6 | 6
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | 9 | 12
Neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 6 | 6
Insomnia (Psychiatric disorders) | 6 | 15 | 8 | 17
Depression (Psychiatric disorders) | 10 | 24 | 11 | 15
Anxiety (Psychiatric disorders) | 3 | 6 | 6 | 8
Headache (Nervous system disorders) | 21 | 42 | 18 | 42
Paraesthesia (Nervous system disorders) | 6 | 26 | 13 | 23
Dizziness (Nervous system disorders) | 5 | 14 | 7 | 14
Hypoaesthesia (Nervous system disorders) | 4 | 20 | 10 | 13
Hypertension (Vascular disorders) | 10 | 22 | 11 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 22 | 7 | 19
Diarrhoea (Gastrointestinal disorders) | 16 | 24 | 19 | 30
Nausea (Gastrointestinal disorders) | 10 | 20 | 10 | 29
Constipation (Gastrointestinal disorders) | 4 | 10 | 7 | 15
Abdominal pain upper (Gastrointestinal disorders) | 3 | 16 | 4 | 10
Abdominal pain (Gastrointestinal disorders) | 5 | 22 | 8 | 9
Toothache (Gastrointestinal disorders) | 2 | 13 | 3 | 9
Vomiting (Gastrointestinal disorders) | 8 | 8 | 5 | 8
Eczema (Skin and subcutaneous tissue disorders) | 2 | 7 | 1 | 15
Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 6 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 12 | 18 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 37 | 16 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 27 | 20 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 31 | 9 | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 1 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 12 | 4 | 13
Micturition urgency (Renal and urinary disorders) | 8 | 4 | 3 | 9
Fatigue (General disorders) | 17 | 37 | 17 | 26
Influenza like illness (General disorders) | 1 | 6 | 1 | 13
Alanine aminotransferase increased (Investigations) | 18 | 36 | 18 | 32
Gamma-glutamyltransferase increased (Investigations) | 4 | 16 | 2 | 12
Aspartate aminotransferase increased (Investigations) | 4 | 18 | 4 | 11
Blood pressure increased (Investigations) | 8 | 10 | 5 | 7
Fall (Injury, poisoning and procedural complications) | 9 | 20 | 8 | 34
Contusion (Injury, poisoning and procedural complications) | 4 | 5 | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.